CLINICAL TRIAL: NCT02041221
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SPARC1316
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPARC_Ltd_ CLR_13_16
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: pharmacokinetics, pharmacodynamics, asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SPARC1316 Dose 1 (Experimental): Subjects will be administered with SPARC1316 dose 1
  Interventions: Drug: SPARC1316 Dose 1
- Placebo (Placebo Comparator): The subjects will receive placebo.
  Interventions: Drug: Placebo
- SPARC1316 Dose 2 (Experimental): Subjects will be administered with SPARC1316 dose 2
  Interventions: Drug: SPARC1316 Dose 2
- SPARC1316 Dose 3 (Experimental): Subjects will be administered with SPARC1316 dose 3
  Interventions: Drug: SPARC1316 Dose 3
- SPARC1316 Dose 4 (Experimental): Subjects will be administered with SPARC1316 dose 4
  Interventions: Drug: SPARC1316 Dose 4
- SPARC1316 Dose 5 (Experimental): Subjects will be administered with SPARC1316 dose 5
  Interventions: Drug: SPARC1316 Dose 5

INTERVENTIONS:
Drug: SPARC1316 Dose 1 — The subjects will receive SPARC1316.
  Arms: SPARC1316 Dose 1
Drug: Placebo
  Other Names: The subjects will receive a matching placebo by oral inhalation.
  Arms: Placebo
Drug: SPARC1316 Dose 2
  Arms: SPARC1316 Dose 2
Drug: SPARC1316 Dose 3
  Arms: SPARC1316 Dose 3
Drug: SPARC1316 Dose 4
  Arms: SPARC1316 Dose 4
Drug: SPARC1316 Dose 5
  Arms: SPARC1316 Dose 5

SUMMARY:
Sun Pharma Advanced Research company Limited has developed a dry powder inhaler of compound SPARC1316 for oral inhalation. This clinical study is a Phase I/IIa study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple ascending doses of S0597 administered by oral inhalation to healthy volunteers and asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to provide informed consent
* Male or female subjects aged 18 to 65 years inclusive
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive
* Non-smokers or ex-smokers

Exclusion Criteria:

* Subjects with a supine systolic blood pressure ≥160 mmHg and/or a supine diastolic blood pressure ≥100 mmHg
* Subjects who have a significant infection or known inflammatory process on screening or admission.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Positive serology for infectious disease (hepatitisB or C , HIV) at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC study site, London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- S0597 Dose 1: Subjects will be administered with SPARC1316 dose 1
- S0597 Dose 2: Subjects will receive SPARC1316 dose 2
- S0597 Dose 3: Subjects will receive SPARC1316 dose 3
- S0597 Dose 4: Subjects will receive SPARC1316 dose 4
- S0597 Dose 5: Subjects will receive SPARC1316 dose 5
- Placebo: Subjects will receive placebo
Period: Part 1
Arm/Group | S0597 Dose 1 | S0597 Dose 2 | S0597 Dose 3 | S0597 Dose 4 | S0597 Dose 5 | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | S0597 Dose 1 | S0597 Dose 2 | S0597 Dose 3 | S0597 Dose 4 | S0597 Dose 5 | Placebo
Started | 6 | 6 | 6 | 0 (Part 1 data fields are by default copied in Part 2. There is no dose 4 and 5 actually.) | 0 (Part 1 data fields are by default copied in Part 2. There is no dose 4 and 5 actually) | 6
Completed | 6 | 6 | 5 | 0 (Part 1 data fields are by default copied in Part 2. There is no dose 4 and 5 actually) | 0 (Part 1 data fields are by default copied in Part 2. There is no dose 4 and 5 actually) | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- S0597 Dose 1: Subjects will be administered with S0597
  S0597: The subjects will receive S0597.
  Placebo
- S0597 Dose 2: The subjects will receive placebo.
  S0597: The subjects will receive S0597.
  Placebo
- Total: Total of all reporting groups
Arm/Group | S0597 Dose 1 | S0597 Dose 2 | S0597 Dose 3 | S0597 Dose 4 | S0597 Dose 5 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Customized [Mean (Standard Deviation); unit: years] | 33 (3.9) | 28 (8.2) | 28 (4.9) | 27 (8.8) | 31 (5.8) | 27 (5.3) | 29 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: The no of adverse events will be assessed to evaluate the safety and tolerability of compound SO597 in healthy male subjects and asthma patients
Time Frame: Two (2) Weeks
Measure: Number; unit: participants
Groups:
- S0597 Dose 1: The subjects will receive placebo.
  S0597: The subjects will receive S0597.
  Placebo
Arm/Group | S0597 Dose 1 | S0597 Dose 2 | S0597 Dose 3 | S0597 Dose 4 | S0597 Dose 5 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
participants | 0 | 0 | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Arm/Group | S0597 Dose 1 | S0597 Dose 2 | S0597 Dose 3 | S0597 Dose 4 | S0597 Dose 5 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S0597 Dose 1 (N=6) | S0597 Dose 2 (N=6) | S0597 Dose 3 (N=6) | S0597 Dose 4 (N=6) | S0597 Dose 5 (N=6) | Placebo (N=10)
URTI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other